CLINICAL TRIAL: NCT01570972
Title: Mediators and Moderators of Treatment Outcome in Recent-Onset Psychosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Nicholas Breitborde, Assistant Professor, Department of Psychiatry, University of Arizona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U. Az IRB 09-1113-02
Record Dates: First submitted 2011-11-07; First posted 2012-04-04 (Estimated); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Bipolar Disorder With Psychotic Features; Major Depression With Psychotic Features; Psychotic Disorder Not Otherwise Specified (NOS)
Keywords: schizophrenia; schizoaffective disorder; bipolar disorder with psychotic features; major depression with psychotic features; recent-onset psychosis; first-episode psychosis; cognitive behavioral therapy; multifamily group psychoeducation
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MFG and GCBT (Other): There is a single arm for this study. All participants will be able to participate in MFG and GCBT
  Interventions: Behavioral: Group Cognitive Behavioral Therapy; Behavioral: Multifamily Group Psychoeducation

INTERVENTIONS:
Behavioral: Group Cognitive Behavioral Therapy — weekly
Behavioral: Multifamily Group Psychoeducation — twice monthly

SUMMARY:
Multifamily group psychoeducation [MFG] and group cognitive behavioral therapy [GCBT] are evidence-based treatments for first episode psychosis. However, like all treatments for psychotic disorders, neither MFG nor GCBT are perfect-some individuals who receive these interventions still experience a worsening of psychotic symptoms. Clarifying the mechanisms through which these interventions produce their clinical benefits and identifying the factors that may maximize an individual's response to MFG and GCBT could improve the clinical benefits facilitated by these two interventions.

DETAILED DESCRIPTION:
Background

There is growing evidence that the majority of the psychosocial deterioration that accompanies psychotic disorders occurs during the first few years of illness and that the prevention or delay of early deterioration may be associated with a better course of illness. Two interventions which have been shown to improve the course of recent-onset psychosis are multifamily group psychoeducation [MFG] and group cognitive behavioral therapy [GCBT]. Both family psychoeducation and cognitive behavioral therapy have been recommended as components of usual care for psychotic disorders by the Schizophrenia Patient Oriented Research Team convened by the U.S. Department of Health and Human Services (10) as well as other international health organizations. However, like all treatments for psychotic disorders, neither MFG nor GCBT are perfect-some individuals who receive these interventions still experience a worsening of psychotic symptoms. Clarifying the mechanisms through which these interventions produce their clinical benefits and identifying the factors that may maximize an individual's response to MFG and GCBT could improve the clinical benefits facilitated by these two interventions.

Purpose and Objectives

The goal of this study is to clarify the mechanisms through which MFG and GCBT produce their clinical benefits (i.e., mediators) and identify the factors that may maximize an individual's response to these two empirically-validated interventions (i.e., moderators).

Methods

All participants will be provided with 2 years of of GCBT and MFG and will complete regular assessments with regard to clinical and functional outcomes as well as potential mediators and moderators of these outcomes.

Significance of the Study

Clarifying the mechanisms through which these interventions produce their clinical benefits and identifying the factors that may maximize an individual's response to MFG and GCBT could lead to improvements in the treatment of first-episode psychosis.

ELIGIBILITY:
Inclusion Criteria (Individual with Recent-Onset Psychosis):

* Diagnosis of a non-substance induced psychotic disorder (schizophrenia spectrum or affective spectrum) per the Diagnostic and Statistical Manual of Mental Disorders-IV-Text Revised (DSM-IV-TR) criteria determined using the Structured Clinical Interview for the DSM-IV.
* Age between 18-35
* Willing to participate in interventions at University of Arizona Medical Center South Campus
* Willing to complete research assessments
* Duration of psychotic symptoms of less than 5 years determined using the Symptom Onset in Schizophrenia inventory
* Able to provide informed consent
* Fluent in English
* Willing to allow videotaping of group cognitive behavioral therapy sessions, multifamily group sessions, and family interaction task.

Exclusion Criterion (Individual with Recent Onset Psychosis)

* No evidence of mental retardation as defined as never having qualified to receive services from the Arizona Department of Economic Security, Division of Developmental Disabilities.

Inclusion Criteria (Family Caregiver):

* Must be someone that the individual with recent-onset psychosis identifies as providing support and care to the individual with recent-onset psychosis. Does not need to be a biological relative.
* Must spend considerable time with the individual with recent-onset psychosis as defined at 10 hours or more of direct contact per week.
* Willing to participate in participate in family intervention at University of Arizona Medical Center, South Campus for 2 years
* Willing to complete research assessments
* Able to provide informed consent
* Fluent in English
* Willing to allow videotaping of multifamily group sessions, Camberwell Family Interview, and family interaction task.

Exclusion Criterion (Family Caregiver)

* Diagnosis of a psychotic disorder.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 103 (Actual)
Dates: Start 2010-02 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in General level of functioning at 6 months, 12 months, 18 months, and 24 months | Baseline, 6 months, 12 months, 18 months, 24 months
  General level of functioning to be assessed using the General Assessment of Functioning (GAF) scale
Change from baseline in self-reported Physical Health at 6 months, 12 months, 18 months, and 24 months | Baseline, 6 months, 12 months, 18 months, 24 months
  Self-reported physical health assessed using the RAND-36 Health Survey
Change from baseline in Social and vocational Functioning at 6 months, 12 months, 18 months, and 24 months | Baseline, 6 months, 12 months, 18 months, 24 months
  Social and Vocational functioning to be assessed using the Social Functioning Scale
Change from baseline in Stage of Recovery at 6 months, 12 months, 18 months, and 24 months | Baseline, 6 months, 12 months, 18 months, 24 months
  Stage of recovery assessed using the Stage of Recovery Instrument
Change from baseline Service Utilization at 6 months, 12 months, 18 months, and 24 months | Baseline, 6 months, 12 months, 18 months, 24 months
  Service utilization as assessed using the Service Utilization Record Form
Change from Baseline Quality of Life at 6 months, 12 months, 18 months, and 24 months | Baseline, 6 months, 12 months, 18 months, 24 months
  Quality of Life as assessed using the WHO Quality of Life Scale Brief

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Breitborde, Ph.D., Principal Investigator — The Ohio State Univerity
Locations (1):
- University of Arizona Department of Psychiatry, Tucson, Arizona, United States

REFERENCES:
- [Derived] Moe AM, Wastler HM, Pine JG, Breitborde NJK. Metacognitive Skills Training and Computerized Cognitive Remediation among Individuals with First-Episode Psychosis: Influence on Social Cognition. Psychosis. 2023;15(4):418-423. doi: 10.1080/17522439.2022.2111595. Epub 2023 Jan 4. PMID 38053744
- [Derived] Breitborde NJK, Bell EK, Woolverton C, Pine JG, Waslter H, Moe AM. Cost Utility of cognition-enhancing interventions for individuals with first-episode psychosis: a naturalistic evaluation. Cost Eff Resour Alloc. 2021 Jul 1;19(1):36. doi: 10.1186/s12962-021-00292-6. PMID 34210341
- [Derived] Breitborde NJ, Bell EK, Dawley D, Woolverton C, Ceaser A, Waters AC, Dawson SC, Bismark AW, Polsinelli AJ, Bartolomeo L, Simmons J, Bernstein B, Harrison-Monroe P. The Early Psychosis Intervention Center (EPICENTER): development and six-month outcomes of an American first-episode psychosis clinical service. BMC Psychiatry. 2015 Oct 28;15:266. doi: 10.1186/s12888-015-0650-3. PMID 26511605